CLINICAL TRIAL: NCT06954454
Title: Impact of In-Person Versus Online Supervised Multicenter Multicomponent Prenatal Exercise Program on Maternal Physical Activity, Fitness, and Healthy Lifestyle - The Active Pregnancy Trial Protocol
Brief Title: Impact of In-Person Versus Online Supervised Multicenter Multicomponent Prenatal Exercise Program on Maternal Physical Activity, Fitness, and Healthy Lifestyle
Acronym: ActivePregnanc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Polytechnic University of Santarém (Other)
Collaborators: SPRINT Sport Physical Activity and Health Research & Innovation Center (Unknown)
Responsible Party: Principal Investigator, Rita Santos-Rocha, Professor, Polytechnic University of Santarém
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023.14896.PEX
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: Pregnant Women Participating in a Supervised Multicomponent Exercise Intervention
Keywords: pregnancy; physical activity; exercise; fitness; women; exercise prescription
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Arm 1: In-Person Exercise Group (IN) Type of exercise: multicomponent prenatal exercise program including aerobic, coordination, strength, stretching, balance, postural, and pelvic floor muscle training exercises.
  Duration and frequency: two sessions of 60 minutes per week for 12 weeks. In-person supervision: qualified exercise physiologists. Setting: healthcare, university, or fitness centers. Arm 2: Online Exercise Group (ON) Type of exercise: multicomponent prenatal exercise program including aerobic, coordination, strength, stretching, balance, postural, and pelvic floor muscle training exercises.
  Duration and frequency: two sessions of 60 minutes per week for 12 weeks. Remote supervision using a virtual platform: qualified exercise physiologists. Setting: home or outdoors. Additional recommendations include educational materials (Active Pregnancy Guide), walking, swimming, or performing a video session from the Active Pregnancy Guide Channel on other days of the week.
Who Masked: Participant, Care Provider
Masking Description: Data analyst are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: In-Person Exercise Group (IN) (Active Comparator): Arm 1: In-Person Exercise Group (IN) Type of exercise: multicomponent prenatal exercise program. Program duration: 12 weeks. Frequency: two weekly sessions. Session duration: 60 minutes. Intensity: moderate. Supervision: qualified exercise physiologists. Setting: healthcare, university, or fitness centers.
  Interventions: Other: prenatal physical exercise intervention
- Arm 2: Online Exercise Group (ON) (Active Comparator): Arm 2: Online Exercise Group (ON) Type of exercise: multicomponent prenatal exercise program. Program duration: 12 weeks. Frequency: two weekly sessions. Session duration: 60 minutes. Intensity: moderate. Supervision: qualified exercise physiologists. Setting: home or outdoors.
  Interventions: Other: prenatal physical exercise intervention

INTERVENTIONS:
Other: prenatal physical exercise intervention — Multicomponent prenatal exercise program including aerobic, coordination, strength, stretching, balance, postural, and pelvic floor muscle training exercises. Delivered either in person or online by qualified exercise physiologists. Duration and frequency: two sessions of 60 minutes per week for 12 weeks. Moderate intensity: According to the Borg scale of perceived exertion, from six to 20, moderate exercise is rated between 13 and 14. Each pregnant woman will rate her exercise on the Borg perceived exertion scale from six to 20. Settings: home or healthcare, university, or fitness centers. Following international guidelines for physical activity during pregnancy (ACOG-USA, ACSM-USA, CSEP-Canada, PSOG-Poland, SEGO-Spain).
  Other Names: physical activity and healthy lifestyle promotion

SUMMARY:
Many studies have been supporting the positive effects of an active lifestyle concerning the prevention and treatment of pregnancy-related complications and health problems, such as gestational diabetes, gestational hypertension, obesity, low back pain, urinary incontinence, anxiety or depression, as well as regarding its effectiveness in maintaining fitness and functionality, and in improving postpartum recovery.

Practice and clinical guidelines have become increasingly popular tools for synthesizing evidence-based information to assist practitioners and patients/participants in making decisions related to starting or continuing physical activity.

Despite this knowledge, most women still do not receive proper guidance on how to exercise during pregnancy or after childbirth, and the prevalence of physical inactivity is still high among pregnant and postpartum women. On the other hand, the COVID-19 pandemic has highlighted the need for virtual approaches in health interventions, but few studies have addressed the effectiveness of such interventions.

This study is about the benefits of exercising during pregnancy in terms of maternal physical activity, fitness, and healthy lifestyle parameters. After the first visit to the doctor, pregnant women without absolute contraindications to exercise will be invited to participate in a multi-site (fitness center, university, or hospital) prenatal exercise program delivered either in person or online by qualified exercise physiologists.

The exercise intervention will follow international evidence-based guidelines. It includes aerobic, coordination, strength, postural, stretching, and pelvic floor exercises, organized in two weekly sessions lasting 60 minutes each.

Pregnant women will be asked to answer questionnaires about physical activity, fitness, and healthy lifestyle parameters (sleep, diet, stress) twice: before starting the exercise program and after completing 12 weeks of the program. The same procedure applies to basic fitness field tests (e.g., to assess balance, flexibility, strength, cardiorespiratory fitness, etc.).

Participants will have access to the free Active Pregnancy Guide (including recommendations for walking, dancing, swimming, etc.). On other days of the week, they can follow specific workouts on the YouTube channel (@GravidezAtiva-ActivePregnancy).

Researchers will test whether the exercise program is beneficial in maintaining or improving maternal physical activity and fitness levels and healthy lifestyle parameters after 12 weeks. Moreover, researchers will compare which exercise mode (in-person or virtual) is better or similar. Participants will also be asked about their satisfaction with the intervention and educational resources. Participation and resources will be free. All participants will benefit from the exercise intervention.

The study's results will contribute to knowledge on this topic, inform future exercise recommendations for pregnant women, and inform public health strategies.

DETAILED DESCRIPTION:
Scientific studies have been supporting the positive effects of an active lifestyle concerning the prevention and treatment of pregnancy-related complications and health problems, such as gestational diabetes, gestational hypertension, obesity, low back pain, urinary incontinence, anxiety or depression, as well as regarding its effectiveness in maintaining fitness and functionality, and in improving postpartum recovery.

Practice and clinical guidelines have become increasingly popular tools for synthesizing evidence-based information to assist practitioners and patients/participants in deciding to start or continue physical activity.

Despite this knowledge, most women still do not receive proper guidance on how to exercise during pregnancy or after childbirth, and the prevalence of physical inactivity is still high among pregnant and postpartum women. On the other hand, the COVID-19 pandemic has highlighted the need for virtual approaches in health interventions, but few studies have addressed the effectiveness of such interventions.

This trial will compare the effectiveness of in-person versus online supervised prenatal exercise programs on improving maternal physical activity, functional fitness, healthy lifestyle parameters, and health outcomes. After the first visit to the doctor, pregnant women without absolute contraindications to exercise will be invited to participate in a multi-site (home, fitness center, university, or hospital) prenatal exercise program delivered either in person or online. The study will be conducted in multiple centers, recruiting women between 13-20 gestational weeks, allocated to in person or online exercise groups for 12 weeks. The exercise intervention will follow international evidence-based guidelines. It includes aerobic, coordination, strength, postural, stretching, and pelvic floor exercises, organized in two weekly sessions lasting 60 minutes each. All sessions will be supervised by qualified exercise physiologists.

Assessments include validated questionnaires (PPAQ, IFIS, etc.) and fitness tests, at baseline and post-intervention. Pregnant women will be asked to answer questionnaires about physical activity (PPAQ), fitness (IFIS), and healthy lifestyle parameters (health, sleep, diet, stress) twice: before starting the exercise program and after completing 12 weeks of the program. The same procedure applies to basic fitness field tests (e.g., to assess balance, flexibility, strength, cardiorespiratory fitness, etc.). All tests will be applied by qualified exercise physiologists.

Demographic data (age, BMI, gestational age) will be described using frequencies and percentages for categorical variables. Descriptive statistics (mean, standard deviation, median, interquartile range) will be used to summarize baseline characteristics of participants in both groups (IN and ON). Descriptive and inferential statistics will be applied to all outcomes. Comparative analysis of IN vs. ON interventions will be conducted using intention-to-treat and per-protocol approaches. Comparative analysis will be used to compare changes in primary (physical activity, health-related, and functional fitness) and secondary (lifestyle parameters) outcomes between IN and ON groups over time (baseline and post-intervention). Subgroup analyses will evaluate potential differences regarding maternal age groups (20-34 years vs. 35-50 years). Adjustments will be performed for potential confounders (e.g., maternal age, baseline fitness levels). The significance level of 0.05 (alpha level) will be set for all statistical tests. Power calculations were performed to ensure the study is adequately powered to detect clinically significant differences between groups. For categorical variables, comparative analysis will be performed using chi-square tests or Fisher's exact tests.

Regarding additional outcome analysis, the evaluation of interventions and resources will be performed by means of descriptive analysis summarizing the usage and satisfaction with resources (Active Pregnancy Guide, Active Pregnancy YouTube channel, and Active Pregnancy app) and satisfaction with exercise interventions.

The statistical software SPSS will be used for data analysis. The study has obtained ethics approval from relevant institutional boards. All participants will be informed about the benefits and objectives of the study. Participation in the exercise programs and assessments is free, and they can leave any time without any consequences. Exercise interventions will be supervised and delivered by qualified exercise physiologists and medical records will be obtained by medical doctors. All educational resources will be available for free. Participant confidentiality will be maintained.

Participants will have access to the free Active Pregnancy Guide (including recommendations for walking, dancing, swimming, etc.). On other days of the week, they can follow specific workouts on the YouTube channel (@GravidezAtiva-ActivePregnancy).

Participants will also be asked about their satisfaction with the intervention and educational resources. Participation and resources will be free. All participants will benefit from the exercise intervention.

The study's results will contribute to knowledge on this topic, inform future exercise recommendations for pregnant women, and inform public health strategies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 13 and 20 gestational weeks at baseline
* Age: 18-50 years
* No absolute contraindications to exercise
* Understand the Portuguese language

Exclusion Criteria:

* Any absolute contraindications to exercise as per guidelines
* High-risk pregnancy conditions requiring physical activity restrictions

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-10-24 (Estimated); Study Completion 2027-04-24 (Estimated)

PRIMARY OUTCOMES:
Physical activity | Baseline (week 0) and after 12-week intervention (week 13)
  Level and pattern of physical activity in type of PA (work, active commuting, exercise, etc.), type of exercise, duration of each session (time spent in PA), weekly frequency, and intensity, weekly volume. Pregnancy Physical Activity Questionnaire (PPAQ) and Get Active Questionnaire for Pregnancy
Self-perceived fitness | Baseline (week 0) and after 12-week intervention (week 13)
  Self-perceived global fitness and fitness components (cardiorespiratory, strength, speed/agility, flexibility) when compared to other women of the same age. Lickert scale 1 (poor) to 5 (very good). IFIS International Fitness Scale
Cardiorespiratory fitness | Baseline (week 0) and after 12-week intervention (week 13)
  Cardiorespiratory fitness - 6-min walk test (average distance covered in m and estimated cardiorespiratory fitness in mL/Kg/min)
Upper limbs strength | Baseline (week 0) and after 12-week intervention (week 13)
  Upper limbs strength - wall push-ups (number of repetitions in 30s)
Lower limbs strength | Baseline (week 0) and after 12-week intervention (week 13)
  Lower limbs strength - sit-and-stand (number of repetitions in 30s)
Dynamic balance | Baseline (week 0) and after 12-week intervention (week 13)
  Dynamic balance - tandem walk.
Static balance | Baseline (week 0) and after 12-week intervention (week 13)
  Static balance - One Leg Stance.
Lower limbs flexibility | Baseline (week 0) and after 12-week intervention (week 13)
  Lower limbs flexibility - modified sit and reach (mm)
Upper limbs flexibility | Baseline (week 0) and after 12-week intervention (week 13)
  Upper limbs flexibility - back scratch (mm).
Agility | Baseline (week 0) and after 12-week intervention (week 13)
  Agility - Time Up & Go over 3 m distance (in min).

SECONDARY OUTCOMES:
Sleep | Baseline (week 0) and after 12-week intervention (week 13)
  Sleep: PSQI Pittsburgh Sleep Quality Index
Weight | Baseline (week 0) and after 12-week intervention (week 13)
  Pre-pregnancy, weight at baseline and weight gain (Kg)
Happiness | Baseline (week 0) and after 12-week intervention (week 13)
  Happiness: SHS Subjective Happiness Scale
Depression | Baseline (week 0) and after 12-week intervention (week 13)
  Depression: EPDS Edinburgh Postpartum Depression Scale.
Diet | Baseline (week 0) and after 12-week intervention (week 13)
  Diet: MEDAS Mediterranean Diet Adherence Screener.
Heart rate | Baseline (week 0) and after 12-week intervention (week 13)
  Rest heart rate (bat/min)
Pregnancy-related symptoms | Baseline (week 0) and after 12-week intervention (week 13)
  Prevalence of pregnancy-related symptoms. Medical records and Get Active Questionnaire for Pregnancy.

OTHER OUTCOMES:
Satisfaction with the intervention | After the intervention (13-14 weeks)
  Participant satisfaction with the intervention and use of educational resources. A questionnaire explicitly made for the intervention evaluating different domains: type of exercises, hardness of the sessions, difficulty in particular exercises, weekly frequency, duration of the sessions, context of intervention (online, outdoor, gym, hospital), satisfaction with the exercise physiologist, satisfaction with the educational resources (Active Pregnancy Guide and YouTube channel), willingness to continue in postpartum, willingness to repeat in future pregnancy, overall satisfaction to be included in the program - Likert scale (1 to 5, being 1 not satisfied at all, and 5 highly satisfied).
Feasibility and adherence | After the intervention (weeks 13-14)
  Feasibility evaluation of the implementation of the exercise program: a) Number of women who declined to participate in the study; b) Number of women who give up participation in the study; c) Adherence to the program (number of days of actual performance of the exercise program while admitted); d) Number of women who completed at least 80% of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Santos-Rocha, Ph.D., Principal Investigator — Polytechnic University of Santarém
Locations (3):
- Portugal (3):
  - School of Medicine - University of Minho, Braga
  - Sport Sciences School of Rio Maior - Polytechnic University of Santarem, Rio Maior
  - Health School of Santarem - Polytechnic University of Santarem, Santarém

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 3 years after the publication of results.
Access Criteria: De-identified data will be shared on request.
URL: https://sprint-sci.com/en/research-innovation/research-projects-external/active-pregnancy-202314896pex

REFERENCES:
- [Background] Santos-Rocha R, Pajaujiene S, Szumilewicz A. ACTIVE PREGNANCY: Workshop on Promotion of Physical Activity in Pregnancy for Exercise Professionals. J Multidiscip Healthc. 2022 Sep 14;15:2077-2089. doi: 10.2147/JMDH.S370453. eCollection 2022. PMID 36128597
- [Background] Santos-Rocha R, Ferreira M, Pimenta N, Branco M, Oviedo-Caro M, Szumilewicz A. Understanding and Involving the Perspective of Pregnant Women as Users When Designing the Framework of e-Health and Exercise Interventions during Pregnancy: Preliminary Study. Healthcare (Basel). 2024 May 30;12(11):1121. doi: 10.3390/healthcare12111121. PMID 38891196
- [Background] Santos-Rocha R, Fernandes de Carvalho M, Prior de Freitas J, Wegrzyk J, Szumilewicz A. Active Pregnancy: A Physical Exercise Program Promoting Fitness and Health during Pregnancy-Development and Validation of a Complex Intervention. Int J Environ Res Public Health. 2022 Apr 18;19(8):4902. doi: 10.3390/ijerph19084902. PMID 35457769
- [Derived] Santos-Rocha R, Branco M, Prior de Freitas J, Castro B, Pinto AT, Silva-Santos S, Nogueira-Silva C, Oviedo-Caro MA, Szablewska A, Szumilewicz A. Impact of in-person versus online supervised multicentre multicomponent prenatal exercise programme on maternal physical activity, fitness and healthy lifestyle: the Active Pregnancy trial SPIRIT 2025-based protocol. BMJ Open Sport Exerc Med. 2025 Jul 11;11(3):e002767. doi: 10.1136/bmjsem-2025-002767. eCollection 2025. PMID 40657545
- See also: Project website — https://sprint-sci.com/pt/investigacao-inovacao/projetos-de-investigacao-externos/gravidez-ativa-202314896pex
- See also: Project YouTube channel — https://www.youtube.com/@gravidezativa-activepregnancy